CLINICAL TRIAL: NCT03938961
Title: Long-stayer Critically Ill Patients: is the Metabolic and Nutritional Therapy in the ICU Creating the Problem?
Brief Title: Metabolic and Nutritional Characteristics of Long-stayer ICU Patients
Acronym: Nutri-ICU-LS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mette M Berger, Clinical Professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER2018-02018
Record Dates: First submitted 2019-04-27; First posted 2019-05-06 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Critically Ill
Keywords: Metabolism, Energy,Glucose, Protein, Energy deficit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intensive care (ICU) patient population has increasing number of very long ICU stays. Long-stayers are usually defined as requiring more than 1 week of mechanical ventilation and of ICU therapy: little is know about their metabolic characteristics and their relation to outcome. The study aims at describing the demographic, nutritional and metabolic aspects of their stay.

Analysis of 200-250 consecutive patients admitted to the ICU long-stayer program.

DETAILED DESCRIPTION:
Data extracted from the computerized ICU system (PDMS): age, Simplified acute physiology score (SAPSII), weight, BMI, Nutrition Risk Score (NRS-2002), daily energy, protein, and glucose intakes, Energy balance, blood glucose (dysglycemia and Glu variability) and lactate, 24hr-insulin (Goal Glu 6-8 mmol/l).

Outcome variables: length of stay (LICU), muscle strength (MRC), vital status at 90 days.

Patients will be followed in detail until ICU discharge and for vital status until day 90 after admission Data will be presented as mean or median, univariate and multivariate analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ICU length of stay > 7 days and enrollment to the long-stayer ICU program

Exclusion Criteria:

* Major burns
* Brain injury
* Severe neurological condition as primary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who required more than 2 weeks of ICU treatment, and who have entered the ICU's long stayer program
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Vital Status | up to 90 days
  Alive or dead at 90 days after ICU admission

SECONDARY OUTCOMES:
Force | up to 90 days
  Muscle strength measured by Medical research Council (MRC) score

OTHER OUTCOMES:
Decubitus ulcer | up to 90 days
  Appearance of decubitus ulcer during ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Adult ICU and Burns, University of Lausanne Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Coded (deidentified) database containing all nutritional, metabolic and laboratory variables

REFERENCES:
- [Background] Loss SH, Nunes DSL, Franzosi OS, Salazar GS, Teixeira C, Vieira SRR. Chronic critical illness: are we saving patients or creating victims? Rev Bras Ter Intensiva. 2017 Jan-Mar;29(1):87-95. doi: 10.5935/0103-507X.20170013. PMID 28444077
- [Result] Viana MV, Pantet O, Bagnoud G, Martinez A, Favre E, Charriere M, Favre D, Eckert P, Berger MM. Metabolic and Nutritional Characteristics of Long-Stay Critically Ill Patients. J Clin Med. 2019 Jul 7;8(7):985. doi: 10.3390/jcm8070985. PMID 31284633